CLINICAL TRIAL: NCT00447655
Title: Improving Outcomes Following Limb Loss: PALS Plus
Acronym: PALS-PLUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC R01DD000153
Record Dates: First submitted 2007-03-14; First posted 2007-03-15 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Amputation
Keywords: Amputation; Self-management; Rehabilitation; Peer support
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Self-management and peer support

SUMMARY:
Limb loss can result from a variety of etiologies including diabetes, trauma and cancer. Following limb loss, individuals are at elevated risk for activity limitations and participation restrictions with significant impact on health and quality of life. Intervention: Working with the Amputee Coalition of America we have developed, evaluated, and established the effectiveness of a self-management program (PALS) to improve health and outcomes following limb loss. Literature suggests that the access to, and effectiveness and utilization of, this class of interventions may be enhanced by the concerted use of early intervention, peer mentorship, motivational interviewing and provider training. Objectives: Our goal is to evaluate the effectiveness of an enhanced, early self-management intervention- PALS Plus. The specific aims are:1) evaluate the effectiveness of the PALS Plus intervention in improving outcomes for persons with limb loss; (2) evaluate the effectiveness of the PALS Plus intervention in maximizing utilization of self-management interventions for persons with limb loss. A cohort of 200 patients will be enrolled prior to implementation of the intervention and will serve as the control group. Subsequently, a second cohort of 200 patients will be enrolled and receive the PALS Plus intervention and will serve as the intervention group. Assessment will be at baseline, treatment completion and six month follow-up. Outcomes: Primary outcome measures are: pain, depressed mood, and positive mood. Secondary outcome measures are: function, participation and bothersomeness of limitations. The investigation will also provide unique and valuable information regarding patients' acceptance and use of peer visitation and self-management following limb loss. Relevance: By establishing the utility and effectiveness of the enhanced self-management intervention, there is the potential to improve the health, activity, participation and quality of life for individuals with disabilities. The intervention addresses the areas of activity and participation in such a way that it can be implemented in local health care facilities working in combination with a national consumer based organization - the Amputee Coalition of America.

DETAILED DESCRIPTION:
Limb loss can result from a variety of etiologies including diabetes, trauma and cancer. Following limb loss, individuals are at elevated risk for activity limitations and participation restrictions with significant impact on health and quality of life. Intervention: Working with the Amputee Coalition of America we have developed, evaluated, and established the effectiveness of a self-management program (PALS) to improve health and outcomes following limb loss. Literature suggests that the access to, and effectiveness and utilization of, this class of interventions may be enhanced by the concerted use of early intervention, peer mentorship, motivational interviewing and provider training. Objectives: Our goal is to evaluate the effectiveness of an enhanced, early self-management intervention- PALS Plus. The specific aims are:1) evaluate the effectiveness of the PALS Plus intervention in improving outcomes for persons with limb loss; (2) evaluate the effectiveness of the PALS Plus intervention in maximizing utilization of self-management interventions for persons with limb loss. Study Design and Participants: The prospective clinical trial will use a two group, lagged-control design to evaluate the intervention at five health care facilities. A cohort of 200 patients will be enrolled prior to implementation of the intervention and will serve as the control group. Subsequently, a second cohort of 200 patients will be enrolled and receive the PALS Plus intervention and will serve as the intervention group. Assessment will be at baseline, treatment completion and six month follow-up. Outcomes: Primary outcome measures are: pain, depressed mood, and positive mood. Secondary outcome measures are: function, participation and bothersomeness of limitations. Improvements in primary and secondary outcomes will result through the impact on self efficacy, patient activation, catastrophizing and social support. The investigation will also provide unique and valuable information regarding patients' acceptance and use of peer visitation and self-management following limb loss. Relevance: By establishing the utility and effectiveness of the enhanced self-management intervention, there is the potential to improve the health, activity, participation and quality of life for individuals with disabilities. The intervention addresses the areas of activity and participation in such a way that it can be implemented in local health care facilities working in combination with a national consumer based organization - the Amputee Coalition of America.

ELIGIBILITY:
Inclusion Criteria:

* Adults (aged 18-85 years) of both sexes and all races admitted to one of the seven participating acute care hospitals or rehabilitation facilities for an amputation procedure and/or treatment immediately following an amputation procedure, including traumatic amputations as well as amputations due to complications for diabetes mellitus, peripheral vascular disease, and malignancy.
* Women and minority patients will be represented in the trial according to the gender and race/ethnic prevalence of patients receiving treatment at the designated hospital and rehabilitation centers.

Exclusion Criteria:

Criteria for exclusion from the study will include:

* Age less than 18 or over 85 years; and
* Inability to communicate in written or spoken English.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2007-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary outcome measures are: pain, depressed mood, and positive mood.

SECONDARY OUTCOMES:
Secondary outcome measures are: function, participation and bothersomeness of limitations

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T Wegener, PHD, Principal Investigator — Johns Hopkins University
Locations (1):
- Good Samaritan Hospital, Baltimore, Maryland, United States